CLINICAL TRIAL: NCT06070103
Title: Depression, Anxiety and Stress Disorders Among Diabetic Patients in Assuit University Hospitals
Brief Title: Depression ,Anxiety and Stress Disorders Among Diabetic Patients in Assuit University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Abdelmoaty Mohamed, resident doctor, Assiut University
Other Study IDs: D,A,S among diabetic Patients
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus
Keywords: depression; anxiety; stress
MeSH Terms: conditions — Diabetes Mellitus; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Assessment the prevalence of psychiatric disorders in diabetic patient in Assuit University Hospital.
2. Determine the associated factors with the psychiatric disorders.

DETAILED DESCRIPTION:
Across the world, both Diabetes and Psychiatric disorders are on rise. Diabetes strongly affects disability, mortality, and global health expenditure. Diabetes mellitus is a disabling long-term health condition that is common and growing. Globally, it affects 10.5% of the population and is the leading cause of lost disability-adjusted life years Type 1 diabetes is a lifelong autoimmune disease characterized by insulin deficiency and resultant hyperglycemia. It constitutes around 10% of all diagnosed cases of diabetes and its incidence is increasing globally. Type 2 diabetes mellitus (DM2) is a chronic metabolic disease characterized by an increase in normal serum glucose levels (hyperglycemia).

Psychological disorders can occur in people with diabetes of all ages. Type 1 diabetes seems to have a higher prevalence of psychological disorders than type 2 diabetes.

About 15%-20% of people with diabetes are suffering from depression. the exact cause of depression in people with diabetes is unknown, it is likely complex due to a combination of genetic, physiological, and psychological factors. Depression and anxiety could worsen the prognosis of diabetes by reducing the patients' ability to self-care and increasing non-compliance to treatments while increasing the risk of serious short-term and long-term complications such as blindness, amputations, stroke, and even premature death.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 70 years Diagnosed according to criteria of the American Diabetes Association fasting plasma glucose (FPG) level of 126 mg/dL (7.0 mmol/L) or higher or A 2-hour plasma glucose level of 200 mg/dL (11.1 mmol/L) or higher during a 75-g oral glucose tolerance test (OGTT).

Exclusion Criteria:

* Patient with cognitive difficulties
* To be very sick and unable to give consent
* Women who were pregnant or had given birth in the last 6 months

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes is a lifelong autoimmune disease characterized by insulin deficiency and resultant hyperglycemia. It constitutes around 10% of all diagnosed cases of diabetes and its incidence is increasing globally. Type 2 diabetes mellitus (DM2) is a chronic metabolic disease characterized by an increase in normal serum glucose levels (hyperglycemia).
Sampling Method: Non-Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression ,Anxiety and stress disorders among diabetic patients in Assuit University Hospitals. | Baseline
  1. Assessment the prevalence of psychiatric disorders in diabetic patient in Assuit University Hospital.
  2. Determine the associated factors with the psychiatric disorders.